CLINICAL TRIAL: NCT00981019
Title: Study of Primary Care Physicians' Understanding and Use of Different Survival Measures
Brief Title: Doctors' Understanding of Survival Statistics
Acronym: MPIB
Status: Completed | Type: Observational
Sponsor: Max Planck Institute for Human Development (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Dr. Odette Wegwarth, Max Planck Institute for Human Development/ Harding Center for Risk Literacy
Other Study IDs: MPIB-01-SM
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-07

CONDITIONS: Screening
Keywords: survival rates; risk communication; screening counselling; screening recommendation; understanding of medical risk

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- mortality*incidence*5-year survival*early stage: Physicians will be faced in scenarios about screening with information on mortality and 5-year survival, followed by information on mortality*incidence and 5-year survival*early stage in a random order.

SUMMARY:
The probably most commonly used measure for expressing the pay-offs of early detection and treatment are survival rates. Yet, over time and groups this metric comes with several biases and thus, is not reliable for judging such benefits. Epidemiologists recommend using reduction of disease-specific mortality rates instead, which is unbiased. The purpose of the study is to investigate how primary care physicians understand and use different survival measures for determining the benefit of cancer screening tests.

ELIGIBILITY:
Inclusion Criteria:

* primary care physicians (internal, general, and family medicine physicians)

Exclusion Criteria:

* all other types of physicians

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 301 primary care physicians (internal, general, and family medicine physicians)
Sampling Method: Non-Probability Sample
Enrollment: 778 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odette Wegwarth, Dr., Principal Investigator — Max Planck Institute for Human Development
Locations (1):
- Max Planck Institute for Human Development, Berlin, Germany

REFERENCES:
- [Derived] Wegwarth O, Schwartz LM, Woloshin S, Gaissmaier W, Gigerenzer G. Do physicians understand cancer screening statistics? A national survey of primary care physicians in the United States. Ann Intern Med. 2012 Mar 6;156(5):340-9. doi: 10.7326/0003-4819-156-5-201203060-00005. PMID 22393129
- See also: Principal investigator's webpage — http://www.mpib-berlin.mpg.de/de/mitarbeiter/odette-wegwarth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sample frame is the Harris Interactive Physician Panel Harris Interactive AG will draw a simple random sample U.S. internal and family medicine physicians from their Physician Panel and e-mail them an invitation and a link to the online-survey
Pre-assignment Details: Inclusion criteria: Physicians in internal, family and general medicine. Exclusion criteria: All physicians other than internal, family and general medicine physicians are excluded from participation because these usually are not offering cancer screening to there patients in the setting of primary care
Groups:
- Mortality*Incidence*5-year Survival*Early Detection Rate: The study-conducted as an online survey study-investigated the influence that different medical statistics such as 5-year survival rates would have on physicians' recommendation behavior for screening and on their judgment of screening's effectiveness. The survey introduced hypothetical scenarios in which a hypothetical patient was requesting a physician's advice on whether to have a screening test. To make that decision the participants (=physicians) were presented with different statistics and then asked if they would recommend the screening to the hypothetical patient and how effective they think the screening would be in reducing cancer mortality. The online survey did not ask any sensitive data.
Period: Overall Study
Arm/Group | Mortality*Incidence*5-year Survival*Early Detection Rate
Started | 778
Completed | 301
Not Completed | 477
Not completed — Did not respond | 65
Not completed — Did not match target population | 94
Not completed — Inadvertent exclusion | 239
Not completed — Hit the survey after closure | 79

BASELINE CHARACTERISTICS:
Arm/Group | Mortality*Incidence*5-year Survival*Early Detection Rate
Number analyzed (Participants) | 778
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 778
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 620
Region of Enrollment [Number; unit: participants]
  United States | 778

OUTCOME MEASURES:

1. Primary Outcome: Number of Physicians (=Participants) Recommending the Screening
Description: The aim of the study was to learn how different medical cancer screening statistics would influence doctors' recommendation behavior and their effectiveness judgments of screening tests. For that reason the online survey study presented physicians with four different medical statistics (e.g., 5-year survival) within four successive scenarios and asked after each scenario whether they would recommend the screening to a (hypothetical) patient given the data. Options to answer are: Definitely yes, Probably yes, Probably no, Definitely no, Can't decide.
Time Frame: 25 minutes (mean duration of the survey)
Population: We calculated that a sample size of 300 physicians was needed to have 90% power to detect differences of 20% or higher in the proportion of respondents correctly answering questions about the different cancer statistics (2-sided alpha of .05).
Measure: Number; unit: participants
Groups:
- Mortality*Incidence*5-year Survival*Early Detection Rate: The survey introduced four different cancer statistics in scenarios about 2 different screening tests. To mask the fact that all statistics stemmed from prostate cancer screening, screening in the scenarios were labeled "X" and "Z". The survey then introduced test Z, whose effectiveness was described in terms of a reduction of cancer mortality. After responding to the series of outcome questions about test Z, physicians received additional information on the cancer incidence, again followed by the outcome questions. In the next scenario, the survey introduced test X, whose effectiveness was described in terms of an increase in 5-year survival and, in the next step, with additional information on early detection rates. After each step, doctors had to respond to the same outcome questions as they had for test Z. Please not, information on test X and test Z were randomly presented to control for order effects.
Arm/Group | Mortality*Incidence*5-year Survival*Early Detection Rate
Number analyzed (Participants) | 301
participants | 301
Statistical Analysis 1: Comparison: Mortality*Incidence*5-year Survival*Early Detection Rate; Study was exploratory, thus no hypotheses had been formalized beforehand. To analyze repeated measures outcomes (e.g., effect of the four different statistic scenarios on doctors' recommendation of screening, their judgment of screening's effectiveness, etc.), we used the McNemar chi-square test and the Wilcoxon signed-rank test. To test for order effects (scenarios were randomly presented)Pearson's chi-square test and the Mann-Whitney U test were used; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Number of Physicians (= Participants) Assuming a Benefit of Screening
Description: Physicians are faced with four different medical statistics about the effect of screening (e.g., 5-year survival) within four successive scenarios and after each scenario asked whether they assume the screening to be beneficial given the statistical information. Options to answer are: yes, no, can't decide. If yes, then participants are further asked to describe this benefit by the following categories: Very large, large, moderate, small, very small.
Time Frame: 25 minutes (mean duration of the survey)
Reporting Status: Not Posted, anticipated posting 2011-08
Measure: Number; unit: participants

ADVERSE EVENTS:
Description: Serious and/or other non-serious adverse events were not collected/not assessed because it was assume that the online survey study, which introduced hypothetical patient cases to doctors, would not results in any adverse events or put the participating doctors at risk.
Arm/Group | Mortality*Incidence*5-year Survival*Early Detection Rate
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Mistaken exclusion of "exclusively outpatient" physicians due to a programming mistake of the online survey screener

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes